CLINICAL TRIAL: NCT07329868
Title: Comparing the Effectiveness of Acceptance and Commitment Therapy and Cognitive Behavioral Stress Management on Fear of Recurrence, Quality of Life, Psychological Distress, and Fatigue of Caregivers of Cancer Patients
Brief Title: Comparison of ACT and CBSM for Caregivers in Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ardakan University (Other)
Responsible Party: Principal Investigator, Fatemeh Al-Sadat Hosseini, Msc Psychology, Ardakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR.YAZD.REC.1403.058
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Caregiver Burden
Keywords: Acceptance and Commitment Therapy; Cognitive Behavioral Sress Management; Fatigue; Quality of Life; Fear of Recurrence; Psychological Distress; Caregivers
MeSH Terms: conditions — Caregiver Burden; Fatigue | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial with three parallel groups. Participants are randomly assigned to one of three groups. The first group receives Cognitive-Behavioral Stress Management (CBSM), the second group receives Acceptance and Commitment Therapy (ACT), and the third group (the control group) receives no intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Behavioral Stress Management (CBSM) (Experimental): Participants in this group receive Cognitive Behavioral Stress Management (CBSM)
  Interventions: Behavioral: Cognitive Behavioral Stress Management (CBSM)
- Acceptance and Commitment Therapy (ACT) (Experimental): Participants in this group receive Acceptance and Commitment Therapy (ACT)
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Control (No Intervention): The control group receives no intervention.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Stress Management (CBSM) — consisted of eight in-person sessions, twice a week for 90 minutes each
  Arms: Cognitive Behavioral Stress Management (CBSM)
Behavioral: Acceptance and Commitment Therapy (ACT) — consisted of eight in-person sessions, twice a week for 90 minutes each
  Arms: Acceptance and Commitment Therapy (ACT)

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of cognitive-behavioral stress management (CBSM) and acceptance and commitment therapy (ACT) on the fear of recurrence, quality of life, psychological distress, and fatigue of caregivers of cancer patients.

Researchers compare the effectiveness of CBSM and ACT to a Control(without receiving intervention) to see if treatment works to improve the health of caregivers of cancer patients. A comparison between the two treatments was also conducted to determine if there was a difference in their effectiveness.

Participants:

In this study, 66 participants were randomly assigned to one of three groups: the CBSM group, the ACT group, or the control group.

The CBSM and ACT groups each attended eight 90-minute, in-person sessions twice a week.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, caregivers had to be 18 years or older, literate, and provide informed consent. A key requirement was that participants either lived with the patient or visited them at least twice a week.

Exclusion Criteria:

Exclusion criteria were applied to ensure the integrity of the study. Participants were excluded if they missed more than two sessions, were currently receiving other psychological interventions, had a major psychiatric or cognitive disorder that would prevent them from providing informed consent, or if the patient passed away.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-09-22 (Actual)

PRIMARY OUTCOMES:
Fear of Cancer Recurrence Inventory-caregiver (FCRI-c) | assessments at three distinct time points: at baseline (pre-intervention), immediately following the four-week intervention period (post-test), and at a two-month follow-up.
  This scale, developed by Lin et al., (2018), consists of 42 items measured on a 5-point Likert scale, encompassing seven subscales related to triggers, severity, psychological distress, functional impairment, insight, reassurance, and coping Strategy.
Depression Anxiety and Stress (DASS) | assessments at three distinct time points: at baseline (pre-intervention), immediately following the four-week intervention period (post-test), and at a two-month follow-up.
  This scale, developed by Lovibond and Lovibond (1995), consists of 21 items measured on a 4-point Likert scale, encompassing three subscales for depression, anxiety, and stress.
Caregiver Quality of Life-Cancer (CQOLC) | assessments at three distinct time points: at baseline (pre-intervention), immediately following the four-week intervention period (post-test), and at a two-month follow-up.
  This scale, developed by Weitzner et al., (1999), consists of 35 items measured on a 5-point Likert scale, encompassing four subscales for burden, disruptiveness, positive adaptation, and financial concern, along with eight additional items.
Multidimensional Fatigue Inventory (MFI) | assessments at three distinct time points: at baseline (pre-intervention), immediately following the four-week intervention period (post-test), and at a two-month follow-up.
  This scale, developed by Smets et al., (1995), consists of 20 items measured on a 5-point Likert scale, encompassing five subscales: general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Emdadgaran-e Ashura Charity Institute, Yazd, Yazd Province, Iran

IPD SHARING:
Plan to Share IPD: No